CLINICAL TRIAL: NCT00030654
Title: A Phase III Randomized Study of Patients With High Risk, Hormone-Naive Prostate Cancer: Androgen Blockade With 4 Cycles of Immediate Chemotherapy Versus Androgen Blockade With Delayed Chemotherapy
Brief Title: Hormone Therapy Plus Chemotherapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network); SWOG Cancer Research Network (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-P-0014; CDR0000069186; ECOG-RTOG-P-0014; CALGB-RTOG-P-0014; SWOG-RTOG-P-0014
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Docetaxel; Doxorubicin; Estramustine; Flutamide; Ketoconazole; Paclitaxel; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Androgen blockade + immediate chemotherapy (Experimental): Androgen blockade with immediate chemotherapy
  Interventions: Drug: bicalutamide; Drug: docetaxel; Drug: doxorubicin hydrochloride; Drug: estramustine phosphate sodium; Drug: flutamide; Drug: ketoconazole; Drug: paclitaxel; Drug: releasing hormone agonist therapy; Drug: vinblastine sulfate
- Androgen blockade + delayed chemotherapy (Experimental): Androgen blockade with delayed chemotherapy
  Interventions: Drug: bicalutamide; Drug: docetaxel; Drug: doxorubicin hydrochloride; Drug: estramustine phosphate sodium; Drug: flutamide; Drug: ketoconazole; Drug: paclitaxel; Drug: releasing hormone agonist therapy; Drug: vinblastine sulfate

INTERVENTIONS:
Drug: bicalutamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: estramustine phosphate sodium
Drug: flutamide
Drug: ketoconazole
Drug: paclitaxel
Drug: releasing hormone agonist therapy
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as luteinizing hormone-releasing hormone agonist, flutamide, and bicalutamide may stop the adrenal glands from producing androgens. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining hormone therapy with chemotherapy may kill more tumor cells. It is not yet known whether chemotherapy given at the same time as hormone therapy is more effective than chemotherapy given after hormone therapy in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy given at the same time as hormone therapy with that of chemotherapy given after hormone therapy in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with high-risk hormone-naive prostate cancer treated with androgen blockade with concurrent chemotherapy vs delayed chemotherapy.

Secondary

* Compare biochemical control in patients treated with these regimens.
* Determine the toxicity of these regimens in these patients.
* Compare the time to clinical failure, as measured by progression on bone scan or CT scan or a prostate-specific antigen (PSA) doubling time of ≤ 32 weeks, in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior therapy (surgery vs radiotherapy and/or brachytherapy vs both), original combined Gleason score (6 vs 7 vs 8-10), and prior vaccine therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive androgen blockade (AB) comprising a luteinizing-hormone releasing-hormone agonist continuously and oral flutamide or oral bicalutamide once daily for at least 1 month. Within 4 weeks of initiation of AB, patients begin chemotherapy. Patients receive 1, and only 1, of the following chemotherapy regimens:

  * Regimen A: Patients receive oral estramustine 3 times daily on days 1-5 and docetaxel IV on day 3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen B: Patients receive oral estramustine 3 times daily on days 1-5 and paclitaxel IV on days 3, 10, 17, 24, 31, and 38. Treatment repeats every 56 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen C: Patients receive oral ketoconazole 3 times daily on days 1-7, 15-21, and 29-35; doxorubicin IV on days 1, 15, and 29; vinblastine IV on days 8, 22, and 36; and oral estramustine 3 times daily on days 8-14, 22-28, and 36-42. Treatment repeats every 56 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen D: Patients receive oral estramustine 3 times daily on days 1-4 and docetaxel IV over 1 hour on days 3, 10, and 17. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen E: Patients receive docetaxel IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen F: Patients receive docetaxel IV on days 1, 8, and 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen G: With approval from the protocol chair, patients may receive a regimen that has been demonstrated in a published phase II study to have at least a 50% response rate as measured by PSA decrease from baseline over 2 measurements 28 days apart or a decrease in measurable soft tissue disease by 50% in 2 dimensions.
* Arm II: Patients receive AB as in arm I. Patients continue with AB until clinical failure, at which time patients receive chemotherapy as in arm I. Patients who have a response may continue to receive chemotherapy beyond 4 courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,050 patients will be accrued for this study within 4-6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Failed local treatments (surgery and/or radiotherapy and/or brachytherapy) as defined by a rising prostate-specific antigen level of at least 2.0 ng/mL (confirmed by 2 measurements at least 2 weeks apart) and a doubling time of 32 weeks or less
  * No clinical or radiographic evidence of disease
  * Original Gleason score of at least 7 OR Gleason score of 6 with capsular penetration or positive seminal vesicles or lymph nodes
* No metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* No history of bleeding disorders that would contraindicate warfarin, including clotting factor defects

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL
* Blood Urea Nitrogen (BUN) no greater than 1.2 times normal

Cardiovascular:

* No symptomatic heart disease
* No history of myocardial infarction
* No history of thromboembolic events (e.g., deep vein thrombosis, symptomatic cerebrovascular events, or pulmonary embolism)

Other:

* No other major medical or psychiatric illness that would preclude study entry
* No other prior or concurrent invasive malignancy within the past 5 years except superficial skin cancer
* No history of esophageal varices
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 weeks since prior vaccine therapy

Chemotherapy:

* At least 5 years since prior chemotherapy

Endocrine therapy:

* Prior adjuvant or neoadjuvant hormonal therapy of less than 8 months duration allowed
* At least 1 year since prior androgen therapy

Radiotherapy:

* See Disease Characteristics
* At least 5 years since prior radiotherapy to sites other than prostate

Surgery:

* See Disease Characteristics

Other:

* Concurrent warfarin allowed
* Concurrent bisphosphonate therapy initiated prior to or after randomization allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-10; Primary Completion 2005-02-04 (Actual); Study Completion 2005-02-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization to the date of death due to any cause

SECONDARY OUTCOMES:
Biochemical control | From date of randomization to the date of first PSA failure defined as a PSA doubling time <= 32 weeks
Time to Clinical Failure | Time from study entry to positive scan or positive disease evaluation of the pelvis or chest or a PSA doubling time ≤ 32 weeks
Frequency of non-hematologic (>= grade 3), hematologic (grade >=4) and fatal (grade 5) toxicities | From the beginning of treatment to 90 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Pienta, MD, FACP, Study Chair — University of Michigan Rogel Cancer Center; Naomi S. Balzer-Haas, MD, Study Chair — Fox Chase Cancer Center; Arif Hussain, MD, Study Chair — University of Maryland Greenebaum Cancer Center; Gregory P. Swanson, MD, Study Chair — Deaconess Medical Center, Spokane, Washington; Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (78):
- United States (75):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - Medical Center of Aurora - South Campus, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers - Denver Rose, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Cancer Research for the Ozarks, Springfield, Missouri
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Akron General's McDowell Cancer Center, Akron, Ohio
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Erlanger Cancer Center, Chattanooga, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Background] Sandler HM, Pienta KJ. Rationale for the Radiation Therapy Oncology Group Study RTOG P-0014. Rev Urol. 2003;5 Suppl 2(Suppl 2):S28-34. PMID 16986043